CLINICAL TRIAL: NCT02310139
Title: Outcomes of Patients With Failed or Difficult Colonoscopy at a Tertiary Referral Centre
Brief Title: Failed/Difficult Colonoscopy Outcomes
Acronym: FoDCO
Status: Completed | Type: Observational
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Other Study IDs: HREC2014/9/4.7(4082)
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Failed/Difficult Colonoscopy: Patients referred for colonoscopy because of previously failed attempt at complete caecal intubation.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy

SUMMARY:
Colonoscopy is a commonly used investigation to diagnose and treat various gastrointestinal disorders. In addition, colonoscopy provides the opportunity to remove colonic adenomas this removal is also known as polypectomy.

Polypectomy has proven to reduce occurrence of colorectal cancer and likelihood of dying from it. Colonoscopy can be challenging due to technical or patient factors. In a small proportion of patients a complete colonoscopy is unsuccessful. Such patients either get referred to a tertiary centre with extensive experience in difficult colonoscopy or have an alternative test such as CT scan. The investigators unit has accumulated significant experience related to previously failed colonoscopy and anecdotally appears to have a high success rate in completing the procedure.

The purpose of this project is to describe the investigators technical approach to management of patients with previously failed colonoscopy. There is no additional intervention and the project is observational in nature. The investigators will collect data on patient characteristics, the reason for the failure and what technique was used to overcome the difficulty. The investigators will also note whether the final outcome of the technique had any impact on the overall management of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Previously failed colonoscopy
* Referred to Westmead Endoscopy Unit for a complete colonoscopy
* 18 years or older

Exclusion Criteria:

* Younger than 18 years
* Previously successful colonoscopy
* No previous colonoscopy attempted

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For a small proportion of patients a complete colonoscopy is unsuccessful due to technical and physical reasons. This will be the study population which will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-05; Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Description of reasons for failure of colonoscopy. | 60 days
  Listing and making note of techniques used to perform successful and complete colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bourke, MBBS, Principal Investigator — Western Sydney Local Health District
Locations (1):
- Westmead Hospital Endoscopy Unit, Sydney, New South Wales, Australia